CLINICAL TRIAL: NCT05044871
Title: The Efficiency of Biomarker-driven Targeted Therapy in Patients With Recurrent Platinum-resistant Epithelial Ovarian Cancer (PROC): An Umbrella Study
Brief Title: Biomarker-driven Targeted Therapy in Patients With Recurrent Platinum-resistant Epithelial Ovarian Cancer
Acronym: BRIGHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Hubei Cancer Hospital (Other); Union Hospital, Tongji Medical College (Unknown); Peking University Cancer Hospital & Institute (Other); Anhui Provincial Hospital (Other Government); Sun Yat-sen University Cancer Center (SUSUCC) (Unknown); Shandong Cancer Hospital and Institute (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Fujian Cancer Hospital (Other Government); Chongqing University Cancer Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-TJ-PROC
Record Dates: First submitted 2021-09-09; First posted 2021-09-16 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer
Keywords: Biomarker-driven; Targeted therapy; Immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pamiparib; Bevacizumab; tislelizumab; Taxes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Pamiparib+ Bevacizumab (Experimental): Arm1 (Biomarkers: BRCA 1/2 mutant): Pamiparib 40mg PO. bid. plus Bevacizumab 7.5mg/kg IV. D1 (q3w.).
  Interventions: Drug: Pamiparib; Drug: Bevacizumab
- Arm 2: Tislelizumab + Bevacizumab + Nab-paclitaxel (Experimental): Arm2 (Biomarkers: BRCA 1/2 wildtype and ≥3 CD8+ TILs count): Tislelizumab 200mg IV. D1 + Bevacizumab 7.5mg/kg IV. D1 + Nab-paclitaxel 125mg / m2 IV. D1, 8 (q3w).
  Interventions: Drug: Bevacizumab; Drug: Tislelizumab; Drug: Nab paclitaxel
- Arm 3: Bevacizumab + Nab-paclitaxel (Experimental): Arm3 (Biomarkers: BRCA 1/2 wildtype and <3 CD8+ TILs count): Bevacizumab 7.5mg/kg IV D1, 15 + Nab-paclitaxel 100mg / m2 IV D1, 8, 15 (Q4w).
  Interventions: Drug: Bevacizumab + Nab paclitaxel (intense dose-dense)

INTERVENTIONS:
Drug: Pamiparib — 40mg PO. bid.
  Arms: Arm 1: Pamiparib+ Bevacizumab
Drug: Bevacizumab — 7.5mg/kg IV. D1 (q3w.)
  Arms: Arm 1: Pamiparib+ Bevacizumab; Arm 2: Tislelizumab + Bevacizumab + Nab-paclitaxel
Drug: Tislelizumab — 200mg IV. D1
  Arms: Arm 2: Tislelizumab + Bevacizumab + Nab-paclitaxel
Drug: Nab paclitaxel — 125mg / m2 IV. D1, 8 (q3w).
  Arms: Arm 2: Tislelizumab + Bevacizumab + Nab-paclitaxel
Drug: Bevacizumab + Nab paclitaxel (intense dose-dense) — Bevacizumab 7.5mg/kg IV. D1, 15 (Q4w). + Nab paclitaxel 100mg / m2 IV. D1, 8, 15 (Q4w).
  Arms: Arm 3: Bevacizumab + Nab-paclitaxel

SUMMARY:
This study is an open-label, multicenter, umbrella study aimed to evaluate the combined, biomarker-driven, targeted treatment efficiency of Pamiparib, Bevacizumab, Tislelizumab, and Nab-paclitaxel in patients with platinum-resistant recurrent ovarian cancer (PROC).

DETAILED DESCRIPTION:
BRCA1/2 gene status and CD8+ tumor-infiltrating T cell count (CD8 + TILs count) were evaluated as biomarkers using archived tumor tissue samples. Treatment arms were arranged according to pathological diagnosis and biomarker detection results.

Arm1 (Biomarkers: BRCA 1/2 mutant): Pamiparib 40mg PO. bid. plus Bevacizumab 7.5mg/kg IV. D1 (q3w.).

Arm2 (Biomarkers: BRCA 1/2 wildtype and ≥3 CD8+ TILs count): Tislelizumab 200mg IV. D1 + Bevacizumab 7.5mg/kg IV. D1 + Nab-paclitaxel 125mg / m2 IV. D1, 8 (q3w).

Arm3 (Biomarkers: BRCA 1/2 wildtype and <3 CD8+ TILs count): Bevacizumab 7.5mg/kg IV D1, 15 + Nab-paclitaxel 100mg / m2 IV D1, 8, 15 (Q4w).

Treatment would continue until disease progression, intolerable toxicity, death, withdrawal of consent, or sponsor termination of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signing of informed consent
2. Age ≥ 18 years;
3. the Eastern United States cancer cooperation group (ECoG) score 0-1;
4. Platinum-resistant recurrent ovarian cancer (PROC): the patient was diagnosed with platinum-resistant recurrence for the first time. PROC refers to the disease progression that occurred < 6 months after the last dose of platinum-based chemotherapy. Imaging-based evaluation for the latest recurrence/progression before enrollment was required;
5. Malignant epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer confirmed by histology or cytology, including high-grade serous cancer, low-grade serous cancer, endometrioid cancer, clear cell cancer, mucinous cancer, and carcinosarcoma;
6. Biomarker detection and tumor sample collection meet the following standards:

   * Patients must provide archived tumor tissue samples (formalin-fixed, paraffin-embedded tumor tissue blocks [preferred], or at least 10 unstained tissue sections), except for patients with serous carcinoma, endometrioid carcinoma, clear cell carcinoma and gBRCAm
   * If the patient has been tested for BRCA1 / 2 gene in the past, only the corresponding test report needs to be provided
7. Sufficient organ functions, which is defined as:

   * neutrophil absolute value (ANC) ≥ 1.5 × 109/L
   * platelet count (PLT) ≥ 75 × 10*9/L
   * hemoglobin ≥ 9 g / dl
   * serum creatinine CR < 1.5 × Upper normal value (ULN)
   * total serum bilirubin ≤ 1.5 × Upper normal range (ULN)
   * both aspartate aminotransferase and alanine aminotransferase ≤ 3 × ULN
   * coagulation function: international normalized ratio (INR) ≤ 1.5; Activated partial prothrombin time (APTT) ≤ 1.5 × ULN
8. Patients must have lesions that can be measured according to RECIST v1.1 standard;
9. Participants were allowed to have previously VEGF / VEGFR inhibitors treatment;
10. Participants were allowed to have previously PARP inhibitors treatment. However, for treatment arm 1 (arm1), the exposure time of PARP inhibitors should ≥ 12 months after first-line chemotherapy or ≥ 6 months after second-line and above chemotherapy;
11. Life expectancy ≥ 3 months;

Exclusion Criteria:

1. The exclusion criteria of bevacizumab were clinically significant cardiovascular and cerebrovascular diseases, history of abdominal fistula or gastrointestinal perforation, acute intestinal obstruction or sub obstruction, and active bleeding;
2. Uncontrolled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) or clinically significant (active) cardiovascular disease: cerebrovascular accident (CVA) / stroke ≤ 6 months from the treatment of the first clinical study; Myocardial infarction ≤ 6 months from the first clinical study treatment; Unstable angina pectoris; Congestive heart failure (CHF) of grade II or above in the cardiac function classification standard of the New York Heart Association (NYHA); Serious arrhythmias requiring treatment;
3. Previous medical history showed newly discovered thrombotic diseases within 6 months before or during the screening period; Patients with severe wound nonunion, ulcer, or fracture;
4. Major surgery within 30 days before the first administration of study treatment; Patients expected to have invasive surgery during treatment;
5. Patients with other malignant tumors;
6. Patients who have previously received anti-programmed cell death protein-1 (anti-PD-1), anti-programmed death ligand-1 (anti-PD-L1) or anti-PD-L2 drugs, or another drug treatment for T cell inhibitory receptors (e.g., cytotoxic T lymphocyte-associated antigen-4 [CTLA-4], OX-40, CD137 [tumor necrosis factor receptor superfamily member 9 (tnfrsf9)];
7. Active autoimmune diseases requiring systemic treatment in the past 2 years;
8. Any case requiring systemic treatment with corticosteroids (prednisone or equivalent > 10 mg/day) or other immunosuppressive drugs ≤ 14 days before the first administration of the study drug;
9. Known history of human immunodeficiency virus (HIV) infection;
10. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA > 500 IU / ml) or active HCV carriers with detectable HCV RNA; Note: inactive hepatitis B surface antigen (HBsAg) carriers and treated and stable hepatitis B patients (HBV DNA < 500 IU / ml) can be included in the group;
11. History of interstitial lung disease, noninfectious pneumonia, or uncontrolled diseases, including pulmonary fibrosis, acute lung disease, etc;
12. Previous heterologous stem cell transplantation or organ transplantation;
13. Peripheral neuropathy ≥ grade 2;
14. Foods or drugs that are expected to use CYP3A4 strong inducers or strong inhibitors within 28 days before the use of the study drug;
15. Participate in another clinical study at the same time, unless it is an observational (non-intervention) clinical study or is in the follow-up period of intervention study;
16. Women of childbearing age who are unwilling or unable to use effective methods for contraception during the whole treatment period of this trial and within 6 months after the last administration of the study drug [women of childbearing age include: any women who have had menarche and have not undergone successful artificial sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or premenopausal], pregnant or lactating women.
17. Other conditions judged by the researcher that do not meet the enrollment requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 108 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR is defined as the proportion of patients with complete response(CR) and partial response(PR) assessed by the investigator in accordance with the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
  PFS is defined as the time from enrollment to the first imaging disease progression or death (whichever occurs first). Assessed according to RECIST v1.1 by investigator.
Overall survival (OS) | Up to 5 years
  OS is defined as the time between enrollment and the patient's death due to any cause.
Disease control rate (DCR) | Up to 5 years
  DCR is defined as the proportion of the patients with complete response, partial remission, and stable disease after treatment. Assessed according to RECIST v1.1 by investigator.
Duration of remission (DOR) | Up to 3 years
  DOR is defined as the time interval from the first record of disease response to disease progression or death (whichever occurs first). Assessed according to RECIST v1.1 by investigator.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 5 years
  Safety includes the adverse event profile of all drugs included according to the Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, MD. PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu Y, Xiong F, Li H, Zheng H, Jiang J, Li Q, Li G, Zhao W, Li R, Li J, Xie R, An R, Zhang H, Gao Q. Biomarker-driven targeted therapy in patients with recurrent platinum-resistant epithelial ovarian cancer (BRIGHT): protocol for an open-label, multicenter, umbrella study. Int J Gynecol Cancer. 2024 Sep 2;34(9):1461-1465. doi: 10.1136/ijgc-2024-005351. PMID 38658024